CLINICAL TRIAL: NCT06766318
Title: Cryo-ultrasound Versus LASER Therapy on Ankle Sprain in Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, Assistant professor, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: REC/012/005532
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Ankle (Ligaments); Instability (Old Injury)
Keywords: cryoultrasound; laser; Ankle sprain; Tennis players; Elite girl
MeSH Terms: conditions — Ankle Injuries | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryo-ultrasound group (n = 20): received cryo-ultrasound therapy (Experimental): received cryo-ultrasound therapy combined with conventional physical therapy
  Interventions: Device: group A will receive cryo-ultrasound therapy combined with conventional physical therapy for two months
- Laser group (Experimental): receive LASER therapy combined with conventional physical therapy
  Interventions: Device: LASER therapy

INTERVENTIONS:
Device: group A will receive cryo-ultrasound therapy combined with conventional physical therapy for two months — Cryo-ultrasound therapy combines two therapeutic methods: cryotherapy (using cold) and ultrasound (using sound waves). The ultrasound component provides a therapeutic heating effect, improving blood circulation and tissue flexibility, while the cold component reduces pain and inflammation
  Arms: cryo-ultrasound group (n = 20): received cryo-ultrasound therapy
Device: LASER therapy — group B will receive LASER therapy combined with conventional physical therapy.
  Arms: Laser group

SUMMARY:
the effect cryo-ultrasound therapy and LASER therapy on the short-term recovery of tennis players with acute lateral ankle sprains.

DETAILED DESCRIPTION:
Acute lateral ankle sprains are common injuries among athletes, but the optimal treatment strategies in elite athletes are still debated. This proof-of-concept study aimed to assess the impact of cryo-ultrasound therapy and LASER therapy on the short-term recovery of tennis players with acute lateral ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 12-16 years.
* elite girls;
* semi-professional tennis players;
* I-II grade lateral ankle sprain injury;
* no persistent instability phenomena or chronic sprains;
* acute injury (within 2 weeks from trauma);
* no evidence of bone edema or skin disorder, once the area of intense pain in motion was delimited, the lack of neurological disturbances was investigated and assessed.

Exclusion Criteria:

* history of recurrent dislocation of the ankle or hyperlaxity of any joint;
* severe rheumatic diseases and/or collagen diseases;
* athletes who have received any form of local physical therapy and NSAIDs within the last 2 months prior to injury;
* athletes who admit to using steroids;
* any contraindication and/or limitation to the use of a physical agent modality (implantable electrophysiological devices, active neoplasms). Taking medications.
* Athletic adult.

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Pain intensity a | 2 months
  We will assess pain intensity before and after intervension by numeric pain rating scale, which is numerical from 0 indicate no pain and 10 indicate the worest pain
Foot and Ankle Disability Index | 2 months
  Foot and Ankle Disability Index (FADI) at baseline (T0) at the end of treatment (T1), after one month (T2), and two months after treatment (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Kerolous Ishak Kelini, PHD, Principal Investigator — AL-Zaytoonah University
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Kerolous Ishak Shehata Kelini, Cairo

IPD SHARING:
Plan to Share IPD: No